CLINICAL TRIAL: NCT01678001
Title: Treatment of Plantar Fasciitis With Xeomin: A Randomized, Placebo-Controlled, Double-Blinded, Prospective Study
Brief Title: Treatment of Plantar Fasciitis With Xeomin
Acronym: Xeomin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Principal Investigator, Jamal Ahmad, Assistant Professor of Orthopaedic Surgery, Rothman Institute Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ IIT - 2011 - 009
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Plantar Fascitis
Keywords: plantar fascia; plantar fascitis; botulinum toxin; Xeomin
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xeomin (Active Comparator): Group A will consist of 25 patients that receive Xeomin. Group B will contain the other 25 patients that receive the placebo saline solution. Post-injection treatment will be kept the same between the two groups. This will only consist of plantar fascial stretching done 3 times daily.
  Interventions: Drug: Xeomin
- Placebo (Placebo Comparator): Group B will contain the other 25 patients that receive the placebo saline solution. Post-injection treatment will be kept the same between the two groups. This will only consist of plantar fascial stretching done 3 times daily.
  Interventions: Drug: Xeomin

INTERVENTIONS:
Drug: Xeomin — Group A will consist of 25 patients that receive Xeomin. Group B will contain the other 25 patients that receive the placebo saline solution. Post-injection treatment will be kept the same between the two groups. This will only consist of plantar fascial stretching done 3 times daily.

SUMMARY:
The plantar fascia is an inelastic, broad band of tissue on the plantar or undersurface of the foot.

Plantar fasciitis is an inflammation of the plantar fascia that causes heel and foot pain.

The current standard orthopaedic management of plantar fasciitis begins with nonsurgical treatment modalities. Surgical treatment of plantar fasciitis is indicated only if nonsurgical means fail.

A newer method of treating plantar fasciitis before resorting to surgery is the use of Botulinum Toxin or Xeomin (incobotulinum toxin A, Merz USA). Treatment of plantar fasciitis with Xeomin is important, as there are limited studies on the subject to date. The purpose of this study is to examine the long-term results of using Xeomin to treat plantar fasciitis in one physician's (J.A.) practice at Rothman Institute Orthopaedics through a placebo-controlled, randomized, double-blinded study.

DETAILED DESCRIPTION:
The plantar fascia is an inelastic, broad band of muscle on the plantar or undersurface of the foot. It runs from the plantar surface of the calcaneus or heel bone to the plantar surface of all 5 toes. The plantar fascia maintains the arch shape of the plantar foot. It also helps with shock absorption upon weight bearing activities such as walking and running.

Plantar fasciitis is an inflammation of the plantar fascia that causes heel and foot pain. This inflammation is often caused by over activity, improper shoes, flat feet, or excessive weight on the feet.

The current standard orthopaedic management of plantar fasciitis begins with nonsurgical treatment modalities. Such methods include daily stretching of the fascia, foot orthotics or inserts to provide arch support, night splinting, and shock-wave therapy. Surgical treatment of plantar fasciitis is indicated only if nonsurgical means fail. However, surgery does have risks, which include but are not limited to bleeding, infection, and nerve injury.

A newer method of treating plantar fasciitis before resorting to surgery is the use of Botulinum Toxin or Xeomin (incobotulinum toxin A, Merz USA). Xeomin can only be delivered via direct injection into the targeted muscle. It takes effect in 2 to 3 days and generally lasts up to 3 to 6 months. Some doctors give Xeomin injections every 3 months or longer for treating spastic muscles. However, others provide single injections to help achieve a specific goal.

Treatment of plantar fasciitis with Xeomin is important, as there are limited studies on the subject to date. Much of the existing research involves BoTox A and non-controlled studies with less than 1 year of patient follow-up. To date, there is only 1 placebo-controlled, randomized, double-blinded study regarding BoTox A to treat plantar fasciitis. However, this study limits its follow-up to 8 weeks. The purpose of this study is to examine the long-term results of using Xeomin to treat plantar fasciitis in one physician's (J.A.) practice at Rothman Institute Orthopaedics through a placebo-controlled, randomized, double-blinded study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be adults above the age of 18 years of any gender or race.
2. Subjects' diagnosis will be plantar fasciitis.
3. Subjects should have attempted 6 weeks of nonsurgical treatment and failed prior to injection.

Exclusion Criteria:

1. Subjects must not have a normal plantar fascia.
2. Subjects must not have received previous BoTox injections at their plantar fascia.
3. Subjects must have not have received prior surgery on their plantar fascia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Function | 1 year
  Function will be scored primarily according to the Foot and Ankle Ability Measure (FAAM), which is validated and reproducible. Scores are based on standing, walking, and performing activities of daily living (ADLs). The scores are between 0 points for being completely disabled and 100 points for being totally without symptoms. A score of 90 or more indicates an excellent result. The PI will gather scores before and after injection. These FAAM scores will be gathered at the time of outpatient follow-up and used to evaluate the final outcome.

SECONDARY OUTCOMES:
Pain | 1 year
  Patients' pain will be scored with a 10 cm visual analog scale (VAS). If applicable, progression to surgical treatment will also be documented.

OTHER OUTCOMES:
Satisfaction | 1 year
  Patients will be asked about their satisfaction by using a CGI satisfaction scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Ahmad, M.D., Principal Investigator — Rothman Institute Orthopaedics
Locations (1):
- Rothman Institute Orthopaedics, Philadelphia, Pennsylvania, United States